CLINICAL TRIAL: NCT02189174
Title: A Phase I/II Multicenter, Open-label Study of CLR457, Administered Orally in Adult Patients With Advanced Solid Malignancies
Brief Title: Study of CLR457 Administered Orally in Adult Patients With Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Novartis decided to terminate the study considering safety and tolerability concerns and limited clinical activity with CLR457 study drug administered once daily (qd).
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCLR457X2101
Record Dates: First submitted 2014-07-07; First posted 2014-07-14 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Advanced Solid Tumor
Keywords: Solid tumor,; breast cancer,; lung cancer,; endometrial cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Endometrial Neoplasms | interventions — CLR457

STUDY DESIGN:
Intervention Model Description: Phase ll part of the study was not conducted as Novartis decided to terminate the study considering safety and tolerability concerns and limited clinical activity.
Oversight: Data Monitoring Committee: No

ARMS (1):
- CLR457 (Experimental)
  Interventions: Drug: CLR457

INTERVENTIONS:
Drug: CLR457

SUMMARY:
To estimate the maximum tolerated dose (MTD) or recommended dose for phase II (RP2D) of CLR457 and to investigate the anti-tumor activity of CLR457

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any screening procedures
* Phase I: Patients with advanced/metastatic solid tumors, with measurable or non-measurable disease as determined by modified RECIST version 1.1 who have progressed despite standard therapy or be intolerant of standard therapy, or for whom no standard therapy exists, who have tumors harboring one of the following: confirmed PIK3CA mutation or amplification, PTEN loss of function, EGFR mutation, cMET activation and/or HER2 overexpression. Endometrial carcinoma will not be selected for any molecular status.
* Phase II: Patients with advanced/metastatic solid tumors, with at least one measurable lesion as determined by modified RECIST version 1.1, who progressed despite standard therapy or be intolerant of standard therapy, or for whom no standard therapy exists, fitting in one of the following groups: Group 1: patients with PIK3CA mutated or amplified ER positive (ER+) breast cancer ; Group 2: patients with endometrial carcinoma (not selected for any molecular status); Group 3: patients with solid tumors (with the exception of PIK3CA mutant/amplified ER+ breast cancer and endometrial carcinoma) harboring PIK3CA mutation or amplification/any PTEN status; Group 4: patients with solid tumors (with the exception of endometrial carcinoma) harboring PTEN loss of function/ PIK3CA wild type; Group 5: non-small cell lung cancer harboring cMET activation and/or EGFR mutation. Up to 3 lines of chemotherapy allowed in advanced/metastatic setting.
* ECOG Performance Status ≤ 2.
* Availability of a representative formalin fixed paraffin embedded tumor tissue sample. If archival tumor sample is not available, a newly obtained tumor sample needs to be submitted instead.

Exclusion Criteria:

* Brain metastasis unless treated and neurologically stable
* Patient having out of range laboratory values defined as:

Hepatic and renal function:

* Serum total Bilirubin ≥ 1.5 x ULN (upper limit of normal) or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2.5 x ULN
* For patients with tumor involvement of the liver AST or ALT > 5 x ULN
* For patients with Gilbert's syndrome total bilirubin > 2.5 x ULN
* Serum creatinine > 1.5 x ULN and/or measured or calculated creatinine clearance < 75% LLN (lower limit of normal)

Bone marrow function:

* Platelets < 100 x 109/L
* Hemoglobin (Hgb) < 9 g/dL
* Absolute Neutrophil Count (ANC) < 1.5 x 109/L

Cardiac function:

* Clinically significant and/or uncontrolled heart disease such as congestive heart failure (CHF) requiring treatment (NYH grade ≥2), hypertension or arrhythmia
* Left ventricular ejection fraction (LVEF) < 45% as determined by MUGA scan or ECHO
* QTcF >480 msec on screening ECG or congenital long QT syndrome
* Acute myocardial infarction (AMI) or unstable angina pectoris < 3 months prior to study entry

  * Peripheral neuropathy CTCAE Grade ≥2
  * History of pancreatitis of any grade
  * Patients with diabetes mellitus requiring insulin treatment and/or with clinical signs or with Fasting Plasma Glucose (FPG) ≥ 140 mg/dL / 7.8 mmol/L
  * Patients receiving treatment with medications that are known to be 1) strong inhibitors or inducers of CYP3A4/5; 2) CYP2C9 substrate with narrow therapeutic index; 3) QT prolonging agents; 4) proton pump inhibitors unless these medications can be discontinued at least a week prior to start of treatment.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-08-07 (Actual); Primary Completion 2015-11-12 (Actual); Study Completion 2015-11-12 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT | First 28 days of dosing
Objective response rate (ORR) as per RECIST v1.1 | Baseline, every 8 weeks until discontinuation for an expected average of 4 months

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Advers Events (SAEs) | Continously throughout the study until 30 days after treatment discontinuation
Severity of AEs and SAEs and dose reductions and interruptions | Continously throughout the study until 30 days after treatment discontinuation
Duration of response (DOR) | Baseline, every 8 weeks until discontinuation for an expected average of 4 months
  per RECIST v1.1
Progression free survival (PFS) | Baseline, every 8 weeks until discontinuation for an expected average of 4 months
  per RECIST v1.1
Best overall response (BOR) | Baseline and every 8 weeks for an expected average of 4 months
  per RECIST v1.1
Plasma concentration and Pharmacokinetics (PK) parameters of CLR457 | During phase I: Baseline; Cycle 1 (C1) Day 1 (D1), 2, 8, 15, 16 and 22; Cycle 2 Day 1, 2, from Cycle 3 to cycle 6 on Day 1 During Phase II: Baseline; Cycle 1 Day 1, 2, 8, 15, 16 and 22
  Parameters including but not limited to Cmax, Cmin, AUCinf, AUCtlast, AUCtau and T1/2
Changes from baseline in glucose metabolism markers (fasting glucose and insulin) | For Phase I and II C1D1, C1D2, C1D15, C1D16 and for Phase I only C2D1 and C2D2
Pre- and post- treatment immunohistochemistry of PI3K pathway molecules in newly obtained paired tumor samples | Baseline, C2D1

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (3):
  - Massachusetts General Hospital SC-9, Boston, Massachusetts
  - Memorial Sloan Kettering SC-4, New York, New York
  - Tennessee Oncology SC, Nashville, Tennessee
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Kashiwa, Chiba, Japan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain